CLINICAL TRIAL: NCT03707483
Title: The Effect of Combination of Vitamin C and Platelet Rich Fibrin (PRF) Versus Platelet Rich Fibrin Alone on Clinical Attachment Gain in Patients With Stage III Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Effect of Incorporation of Vitamin C Into Platelet Rich Fibrin Scaffold in Treatment of Intra-osseous Periodontal Defects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Talaat Mohamed Mahmoud El Behwashy, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: perio285reg
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2018-10

CONDITIONS: Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 250 μM of vitamin C will be used with the platelet rich fibrin
  Interventions: Combination Product: combination of vitamin C and platelet rich fibrin
- Comparator (Active Comparator): using platelet rich fibrin alone
  Interventions: Combination Product: combination of vitamin C and platelet rich fibrin

INTERVENTIONS:
Combination Product: combination of vitamin C and platelet rich fibrin — combination of vitamin C and platelet rich fibrin

SUMMARY:
This study is meant to assess clinically the possible predictable clinical attachment gain regarding the use of vitamin C with platelet rich fibrin versus platelet rich fibrin alone in the treatment of periodontal intrabony defects

DETAILED DESCRIPTION:
Treatment of intra-osseous defects through incorporation of vitamin C into platelet rich fibrin scaffold aims to enhance the biologic potential of the endogenous mesenchymal stem cells that exist within the periodontal ligaments and stimulate periodontal tissue regeneration(Yan et al., 2013). As the concept of periodontal tissue-engineering has emerged, many inductive biomolecules were investigated for periodontal regeneration(Bartold et al., 2000).

Vitamin C has shown promising results in periodontal regeneration, in a study vitamin C was suggested to enhance osteoblastic differentiation of periodontal ligament cells through modulating type I collagen-α1β2 integrin interaction leading to increased ALP activity in periodontal ligament cells(Ishikawa et al., 2004). Vitamin C treatment induces expression of cementogenic genes and considered to be a more feasible and safer treatment for clinical cell-based periodontal regeneration(Gauthier et al., 2017).

There is also a study concluding that vitamin C induces the osteogenic differentiation of PDL progenitor cells via PELP1-ERK axis; and this implies that vitamin C may have a potential in the periodontal regeneration(Yan et al., 2013).

Periodontal tissue regeneration aims to increase periodontal in intra-osseous defects thus improving clinical attachment level; reducing probing depth and upgrading the prognosis of teeth(Ramseier et al., 2012).

Resolution of intra-osseous defects through regeneration preserves and improves function and provides patient comfort(Wang et al., 2005). It also facilitates supportive periodontal therapy; performed regularly to maintain periodontal health(Ramseier et al., 2012).

ELIGIBILITY:
Inclusion Criteria:

* Patient consulting in the outpatient clinic.
* Able to tolerate surgical periodontal procedures.
* Patient ready to perform oral hygiene instructions.
* Compliance with the maintenance program.
* Provide informed consent.
* Accept the 6 months follow-up period
* Mature permanent tooth.
* Tooth with two or three-walled intra-bony defect, CAL ≥ 5mm with intra-osseous defect ≥ 3mm.

Exclusion Criteria:

* Medically compromised patients.
* Pregnant or nursing women.
* Uncooperative patients.
* Smokers.
* Teeth with one wall intra-bony defect.
* Teeth with supra-bony defects.
* Teeth with grade III mobility.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
gain in clinical attachment level | 6 months
  Measured from the CEJ to the bottom of the gingival sulcus

IPD SHARING:
Plan to Share IPD: Undecided